CLINICAL TRIAL: NCT04173507
Title: A Phase II Study of Talazoparib Plus Avelumab in Patients With Stage IV or Recurrent Non-Squamous Non-Small Cell Lung Cancer Bearing Pathogenic STK11 Genomic Alterations (LUNG-MAP Sub-Study)
Brief Title: Combination Treatment (Talazoparib Plus Avelumab) for Stage IV or Recurrent Non-Squamous Non-Small Cell Lung Cancer With STK11 Gene Mutation (A LUNG-MAP Treatment Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1900C; NCI-2019-07142 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1900C (Other: SWOG); S1900C (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Advanced Lung Non-Squamous Non-Small Cell Carcinoma; Recurrent Lung Non-Squamous Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — avelumab; talazoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talazoparib, avelumab) (Experimental): Patients receive talazoparib PO daily and avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avelumab; Drug: Talazoparib; Drug: Talazoparib Tosylate

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673
Drug: Talazoparib Tosylate — Given PO
  Other Names: Talzenna

SUMMARY:
This phase II LUNG-MAP treatment trial studies how well combination treatment (talazoparib plus avelumab) works in treating patients with non-squamous non-small cell lung cancer that has an STK11 gene mutation and has come back (recurrent) or is stage IV. Talazoparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Immunotherapy drugs given as single therapies or in combination with chemotherapy do not appear to work as well in lung cancer cells with mutations in the STK11 gene versus those that do not have the mutation. Adding the medicine talazoparib to the immunotherapy drug avelumab may work better in treating lung cancers that have an STK11 gene mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate (ORR) (confirmed and unconfirmed, complete and partial) with talazoparib plus avelumab in patients with stage IV or recurrent non-squamous non-small cell lung cancer bearing pathogenic STK11 genomic alterations that were previously-treated with anti-PD-1/PD-L1 therapy and platinum-based chemotherapy.

II. To evaluate disease control rate at 12 weeks (DCR12) after registration.

SECONDARY OBJECTIVES:

I. To evaluate investigator assessed progression-free survival (IA-PFS). II. To evaluate overall survival (OS). III. To evaluate duration of response (DOR) among responders. IV. To evaluate the frequency and severity of toxicities.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To collect, process, and bank cell-free deoxyribonucleic acid (DNA) (cfDNA) at baseline, cycle 3 day 1, progression, and end of treatment for future development of a proposal to evaluate comprehensive next-generation sequencing of circulating tumor DNA (ctDNA) and examine molecular mechanisms of resistance to talazoparib and avelumab.

II. To establish a tissue/blood repository from patients with refractory non-small cell lung cancer (NSCLC).

III. To evaluate clinical outcomes (ORR, IA-PFS, OS) in patients with concurrent somatic mutations in KEAP1 detected on the Foundation Medicine Inc. (FMI) panel from the LUNGMAP screening protocol.

IV. To evaluate clinical outcomes (ORR, IA-PFS, OS) in patients with concurrent mutations in ATM or other DNA damage response genes detected on the FMI panel from the LUNGMAP screening protocol.

V. To evaluate the association between tumor mutational burden (TMB) measured on the FMI panel from the LUNGMAP screening protocol and clinical outcomes (ORR, IA-PFS, OS).

OUTLINE:

Patients receive talazoparib orally (PO) daily and avelumab intravenously (IV) over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up until death or 3 years after sub-study registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be assigned to S1900C. Assignment to S1900C is determined by the LUNGMAP protocol genomic profiling using the FoundationOne assay. Biomarker eligibility for S1900C is based on the identification of a pathogenic somatic mutation in STK11 or STK11 bi-allelic loss on tumor
* Patients must have histologically or cytologically confirmed stage IV or recurrent non-squamous, mixed squamous/non-squamous (e.g., adeno-squamous carcinoma), or non-small cell lung cancer not otherwise specified (NSCLC NOS). Patients with pure squamous cell carcinoma are not eligible
* Patients with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy within 28 days prior to sub-study registration
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with HCV infection who are currently on treatment must have an undetectable HCV viral load within 28 days prior to sub-study registration
* Patients with known human immunodeficiency virus (HIV) infection are eligible, provided they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 6 months prior to sub-study registration
* Patients must have received at least one line of anti-PD-1 or anti-PD-L1 therapy for stage III, IV or recurrent disease. Any number of additional, non-platinum-based chemotherapy or targeted therapy regimens for recurrent or metastatic disease are allowed

  * Patients may not have received more than one line of anti-PD-1 or anti-PD-L1 therapy in the Stage IV or recurrent setting. Anti-PD-1 or anti-PD-L1 therapy may have been given alone or in combination with platinum-based chemotherapy, an anti-CTLA4 therapy, or other immune-modulatory therapy. Patients must have experienced disease progression > 42 days following initiation (cycle 1 day 1) of the anti-PD-1 or anti-PD-L1 containing regimen
  * Patients who did not receive anti-PD-1 or anti-PD-L1 therapy in combination with platinum-based chemotherapy, must have also received prior platinum-based chemotherapy and experienced disease progression > 42 days following initiation (cycle 1 day 1) of platinum based chemotherapy
  * Patients who received anti-PD-1 or anti-PD-L1 therapy following concurrent chemoradiation for stage III disease as their only line of anti-PD-1 or anti-PD-L1 therapy, are eligible if they experienced disease progression less than (<) 365 days from the date of initiation of anti-PD-1 or anti-PD-L1 therapy
* Patients who received prior adjuvant platinum-based therapy post-surgical resection for stage I-III disease (i.e. the patient has not received platinum-based chemotherapy for Stage IV or recurrent disease) must have had disease progression during or after platinum-based chemotherapy that occurred less than (<) 365 days from the last date that the patient received that therapy
* Patients must be able to swallow capsules whole
* Patients must not have had prior exposure to any agent with a PARP inhibitor (e.g., veliparib, olaparib, rucaparib, niraparib, talazoparib) as its primary pharmacology
* Patients must not be taking, nor plan to take while on protocol treatment strong P-glycoprotein (P-gp) inhibitors (e.g. dronedarone, quinidine, ranolazine, itraconazole, ketoconazole), P-gp inducers (rifampin, ritonavir, tipranavir), or strong breast cancer resistance protein (BCRP) inhibitors (e.g. elacridar)
* Patients must have progressed following their most recent line of therapy
* Patients must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 21 days prior to sub-study registration. Patients must have recovered (=< grade 1) from any side effects of prior therapy. Patients must not have received any radiation therapy within 14 days prior to sub-study registration
* Patients must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable
* Patients must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI). The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. Measurable disease must be assessed within 28 days prior to sub-study registration. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to sub-study registration. All disease must be assessed and documented on the Baseline Tumor Assessment Form. Patients whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to sub-study registration. CT and MRI scans must be submitted for central review via Transfer of Images and Data (TRIAD)
* Patients must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to sub-study registration. Patient must not have leptomeningeal disease, spinal cord compression or brain metastases unless: (1) metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days following treatment, and prior to sub-study registration, AND (2) patient has no residual neurological dysfunction and has been off corticosteroids for at least 24 hours prior to sub-study registration
* Patient must not have had a major surgery within 14 days prior to sub-study registration. Patient must have fully recovered from the effects of prior surgery in the opinion of the treating investigator
* Serum bilirubin =< institutional upper limit of normal (IULN) (within 28 days prior to sub-study registration). For patients with liver metastases, bilirubin must be =< 5 x IULN
* Either alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 2 x IULN within 28 days prior to sub-study registration (if both ALT and AST are done, both must be =< 2 IULN). For patients with liver metastases, either ALT or AST must be =< 5 x IULN (if both ALT and AST are done, both must be =< 5 x IULN)
* Patients must have a serum creatinine =< the IULN or calculated creatinine clearance >= 50 mL/min using the following Cockcroft-Gault formula. This specimen must have been drawn and processed within 28 days prior to sub-study registration
* Patients must have Zubrod performance status 0-1 documented within 28 days prior to sub-study registration
* Patients must not have any grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia
* Pre-study history and physical exam must be obtained within 28 days prior to sub-study registration
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Absolute neutrophil count (ANC) >= 1,500/mcl (obtained within 28 days prior to sub-study registration). Patients must be transfusion independent (i.e., no blood product transfusions for a period of at least 14 days prior to sub-study registration)
* Platelet count >= 100,000 mcl (obtained within 28 days prior to sub-study registration). Patients must be transfusion independent (i.e., no blood product transfusions for a period of at least 14 days prior to sub-study registration)
* Hemoglobin >= 9 g/dL (obtained within 28 days prior to sub-study registration). Patients must be transfusion independent (i.e., no blood product transfusions for a period of at least 14 days prior to sub-study registration)
* Patients must agree to have blood specimens submitted for circulating tumor DNA (ctDNA)
* Patients must also be offered participation in banking and in the correlative studies for collection and future use of specimens

Exclusion Criteria:

* Patients must not be pregnant or nursing. Women/men of reproductive potential must have agreed to use an effective contraceptive method. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must not have a history of prior organ transplantation, including allogeneic stem-cell transplantation
* Patients must not have received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 7 days prior to sub-study registration. Inhaled or topical steroids, and adrenal replacement doses =< 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease
* Patients must not have active autoimmune disease that requires systemic steroids (equivalent of > 10 mg of prednisone) or immunosuppressive agents within 7 days prior to sub-study registration (for example disease-modifying anti-rheumatic drugs). Exceptions include: patients with controlled type 1 diabetes mellitus, controlled hypo- or hyperthyroidism, vitiligo, resolved childhood asthma/atopy, or psoriasis not requiring immunosuppressive therapy
* Patients must not have any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of talazoparib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or active peptic ulcer disease). Patients must not have active small or large intestine inflammation such as Crohn's disease or ulcerative colitis within 12 months prior to sub-study registration
* Patients must not have known prior or suspected hypersensitivity to monoclonal antibodies (grade >= 3)
* Patients must not have any history of anaphylaxis or uncontrolled asthma. Uncontrolled asthma is defined as a patient having any one of the following criteria:

  * Poor symptom control: Asthma Control Questionnaire (ACQ) consistently > 1.5 or Asthma Control Test Questionnaire (ACT) < 20 (or "not well controlled" by National Asthma Education and Prevention Program [NAEPP] or Global Initiative for Asthma [GINA] guidelines over the 3 months or evaluation)
  * Frequent severe exacerbations: 2 or more bursts of systemic corticosteroids (CSs) (> 3 days each) in the previous year
  * Serious exacerbations: at least one hospitalization, intensive care unit stay or mechanical ventilation in the previous year
  * Airflow limitation: Forced expiratory volume in 1 second (FEV1) < 80% predicted (in the presence of reduced FEV1/forced vital capacity [FVC] defined as less than the normal lower limit) following a withhold of both short- and long-acting bronchodilators
* Patients must not have experienced any immune related adverse event, including pneumonitis that led to permanent discontinuation of prior immunotherapy and/or required prolonged high dose of steroids
* Patients must not have evidence of active infection requiring systemic therapy
* Patients must not have received any live attenuated vaccinations within 28 days prior to sub-study registration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinandos Skoulidis, Principal Investigator — SWOG Cancer Research Network
Locations (325):
- United States (325):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Genesis Cancer Center - Silvis, Silvis, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Western Maryland Regional Medical Center, Cumberland, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - University of Rochester, Rochester, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Jefferson Healthcare, Port Townsend, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 participants were initially registered. Five participants were ineligible. In all, 42 participants were eligible and received protocol therapy.
Groups:
- Talazoparib Plus Avelumab: Participants receive talazoparib PO daily and avelumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Talazoparib: Given PO Avelumab: Given IV
Period: Overall Study
Arm/Group | Talazoparib Plus Avelumab
Started | 42
Completed | 0
Not Completed | 42
Not completed — On Treatment | 3
Not completed — Adverse Event | 3
Not completed — Progression/Relapse | 34
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Eligible participants
Arm/Group | Talazoparib Plus Avelumab
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 63.8 [36.8 to 83.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Prior Lines of Treatment for Stage IV Disease [Count of Participants; unit: Participants]
  0 | 4
  1 | 16
  2 or more | 22
Performance Status [Count of Participants; unit: Participants] — Participants were graded according to the Zubrod Performance Status Scale. 0 - Fully active, able to carry out on all pre-disease performance without restriction.
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work.
  Participants
    0 | 10
    1 | 32
Weight Loss in the Past 6 Months [Count of Participants; unit: Participants]
  < 5% | 25
  5 - < 10% | 12
  10 - < 20% | 3
  Unknown | 2
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 17
  Former Smoker | 23
  Never Smoker | 2
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 36
  Other non-small cell, NOS | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Percentage of participants with confirmed or unconfirmed, complete or partial response to treatment with talazoparib plus avelumab per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria.
  Complete Response (CR): Complete disappearance of all target and non-target lesions. No new lesions. No disease related symptoms. Any lymph nodes (whether target or non-target) must have reduction in short axis to < 1.0 cm. All disease must be assessed using the same technique as baseline.
  Partial Response (PR): Applies only to participants with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: From date of registration to progression or treatment discontinuation, up to 1 year and 9 months
Population: Eligible and evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talazoparib Plus Avelumab
Number analyzed (Participants) | 42
percentage of participants | 2 [0 to 7]

2. Primary Outcome: Disease Control Rate at 12 Weeks (DCR12)
Description: Percentage of participants with a best response of Complete Response (CR), Partial Response (PR), Unconfirmed Partial Response (UPR), or Unconfirmed Complete Response (UCR) by/at the second disease assessment at 12 weeks after registration (+/- 2 weeks), or stable disease at 12 weeks after registration (+/- 2 weeks). Participants with missing or delayed disease assessment at 12 weeks (+/- 2 weeks), at or before the disease assessment at 20 weeks (+/- 2 weeks) with documented lack of progression (CR, PR, UPR, UCR, or stable) were coded as having disease control at 12 weeks. Participants not known to have disease control at 12 weeks who have at least 12 weeks of follow-up were coded as not having disease control at 12 weeks.
Time Frame: 12 weeks after registration
Population: Eligible and evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talazoparib Plus Avelumab
Number analyzed (Participants) | 42
percentage of participants | 40 [26 to 55]

3. Secondary Outcome: Investigator-Assessed Progression-Free Survival (IA-PFS)
Description: From date of sub-study registration to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause. Participants last known to be alive without report of progression are censored at date of last disease assessment. For participants with a missing scan (or consecutive missing scans) whose subsequent scan determines progression, the expected date of the first missing scan (as defined by the disease assessment schedule) is used as the date of progression.
  Progression is defined as: 20% increase in the sum of appropriate diameters of target lesions and absolute increase of at least 0.5 cm, or unequivocal progression of non-measurable disease, or appearance of any new lesion/site, or death from disease without prior documentation of progression or symptomatic deterioration.
  Symptomatic deterioration: Global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talazoparib Plus Avelumab
Number analyzed (Participants) | 42
months | 2.7 [1.6 to 3.9]

4. Secondary Outcome: Overall Survival (OS)
Description: From date of sub-study registration to date of death due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talazoparib Plus Avelumab
Number analyzed (Participants) | 42
months | 7.6 [6.3 to 12.2]

5. Secondary Outcome: Duration of Response (DOR)
Description: From date of first response to first progression assessed by local review or symptomatic deterioration, or death among patients with a response (CR or PR). Those last known to be alive without progression are censored at date of last disease assessment. For those with a missing scan whose next scan shows progression, expected date of the first missing scan is used as progression date.
  Complete Response (CR): Disappearance of all target and non-target lesions. No new lesions or disease related symptoms. Lymph nodes must have reduction in short axis to < 1.0cm. Assessed using same technique as baseline.
  Partial Response (PR): At least 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. Assessed using same technique as baseline.
  Symptomatic deterioration: Global deterioration of health status requiring discontinuation of treatment w/o objective evidence of progression.
Time Frame: From date of registration to a maximum of 3 years or death
Population: Participant with a complete or partial response. As only one participant achieved a response, outcome data is entered as a single number rather than a median.
Measure: Number; unit: months
Arm/Group | Talazoparib Plus Avelumab
Number analyzed (Participants) | 1
months | 7.3

6. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. CTCAE Version 5.0 was used for routine toxicity reporting and serious adverse events (SAEs).
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Eligible participants who received at least one dose of protocol treatment
Measure: Number; unit: Participants
Arm/Group | Talazoparib Plus Avelumab
Number analyzed (Participants) | 42
Participants
  Anemia | 12
  Anorexia | 1
  Atrial flutter | 1
  Fatigue | 1
  Febrile neutropenia | 1
  Generalized muscle weakness | 1
  Hypokalemia | 1
  Hyponatremia | 1
  Hypoxia | 1
  Lung infection | 2
  Lymphocyte count decreased | 5
  Metabolism and nutrition disorders - Other, specify | 1
  Neutrophil count decreased | 1
  Non-cardiac chest pain | 1
  Pain | 1
  Pain in extremity | 1
  Platelet count decreased | 7
  White blood cell decreased | 2

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow-up until death or 3 years post registration
Description: CTCAE Version 5.0 was used for routine toxicity reporting and Serious Adverse Event (SAE) reporting. 42 participants were assessed for adverse events.
Arm/Group | Talazoparib Plus Avelumab
All-Cause Mortality (participants affected / at risk) | 30/42
Serious Adverse Events (participants affected / at risk) | 15/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib Plus Avelumab (N=42)
Anemia (Blood and lymphatic system disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Disease progression (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Lung infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Nervous system disorders-Other (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib Plus Avelumab (N=42)
Anemia (Blood and lymphatic system disorders) | 25
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 13
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 15
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 8
Chills (General disorders) | 4
Fatigue (General disorders) | 23
Fever (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 9
Infusion related reaction (Injury, poisoning and procedural complications) | 5
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 4
Creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 12
Neutrophil count decreased (Investigations) | 10
Platelet count decreased (Investigations) | 17
Weight loss (Investigations) | 13
White blood cell decreased (Investigations) | 13
Anorexia (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 6
Paresthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT04173507/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT04173507/ICF_001.pdf